CLINICAL TRIAL: NCT04841967
Title: Feasibility and Pilot Testing of the TELL Tool Among Gamete and Embryo Donation Recipient Parents
Brief Title: Feasibility Trial of the TELL Tool Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Patricia Hershberger, PhD, RN, FNP-BC, FAAN, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-1086; R34NR019278 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Fertility Issues; Disclosure; Parenting
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Parent participants will be randomized to one of two groups: (1) TELL Tool group, or (2) eBook attention control group. Data will be collected at baseline, immediate posttest (post-TELL tool/post-eBook attention control) and at 2 additional time points (months 1 and 3)
Who Masked: Participant, Investigator
Masking Description: Parents will be randomized into two groups (either the TELL Tool group or the attention control eBook group) using a permuted block approach that is stratified by the age categories of the parent's children and using an online (REDCap) randomization module.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELL Tool Group (Experimental): Parents in the TELL Tool group will complete a decision support aid that has four interactive, multimedia and multicomponent modules that will be administered digitally. It will take parents about 60 minutes to complete the TELL Tool.
  Interventions: Behavioral: TELL Tool Intervention
- eBook Attention-Control (Active Comparator): Parents in the eBook attention-control group will complete one interactive, multimedia and multicomponent program that contains information about good parenting principles and is administered digitally. It will take parents about 60 minutes to complete the eBook attention control.
  Interventions: Behavioral: eBook Attention Control

INTERVENTIONS:
Behavioral: TELL Tool Intervention — A 60-minute session with decision support information delivered digitally to parents at their homes or other private, quiet location.
  Other Names: TELL Tool
  Arms: TELL Tool Group
Behavioral: eBook Attention Control — A 60-minute session with good parenting principles delivered digitally to parents at their homes or other private, quiet location.
  Other Names: eBook
  Arms: eBook Attention-Control

SUMMARY:
A radical paradigm shift is taking place where technology, notably the explosion in easy accessible direct-to-consumer genetic testing (e.g., 23andMe) and a high consumer interest in genealogy (e.g., Ancestry.com), has hijacked gamete (eggs, sperm) and embryo donation recipient parents' control over whether to inform their children about their donor conception. Historically, the practice of gamete donation has been shrouded in secrecy, however, the skyrocketing use of direct-to-consumer genetic testing means that at any point in an adult life, an uninformed donor-conceived person can learn their DNA does not match their presumed ancestry of their parents and family members, putting into question their genetic relatedness to their parents and launching a spiraling sequence of negative health consequences and trauma. Furthermore, the lack of one's knowledge about actual genetic heritage in the age of precision medicine can be enormously detrimental to health and can result in medical maltreatment, including death. To address this serious problem and in accordance with International Patient Decision Aid Standards, we developed a digital, tailored, multicomponent Tool to Empower ParentaL TeLling and Talking (i.e., TELL Tool). The objective of this R34 study is to examine the feasibility, acceptability, and preliminary effects of the TELL Tool intervention in a pilot randomized-controlled feasibility trial with 60 donor-recipient parents and 10 clinicians to determine intervention viability and inform a larger, efficacy trial. An eBook with content about good parenting principles serves as the attention control.

DETAILED DESCRIPTION:
The feasibility trail will use a longitudinal, mixed-methods design that is guided by International Patient Decision Aid Standards and NIH Guidelines for pilot studies. The study design is necessary to achieve the objective of the study, which is to examine the feasibility and acceptability of the TELL Tool intervention in a pilot randomized-controlled feasibility trial to determine intervention viability and inform a larger, efficacy trial. There are three Specific Aims that are: Aim 1 determine feasibility of the study procedures (e.g., recruitment, retention) by pilot testing the TELL Tool using a 2-arm randomized-controlled trial (RCT) with 60 donor-recipient parents using pre- to post-test measures for disclosure intention, competence, and anxiety. (A pretesting of the measures will be implemented with 8 to 12 donor-recipient parents, who are not participants of the pilot RCT, prior to launching the RCT.); Aim 2 survey participating donor-recipient parents at 2 additional time points (4 and 12 weeks/months 1 and 3) post-intervention/attention control completion to obtain meaningful outcome data about actual parental disclosure to their donor-conceived children; and Aim 3 refine the study tools (e.g., TELL Tool, eBook) through post-intervention/attention control written evaluations with participating donor-recipient parents and cognitive interviews with 10 donor-recipient parents, who are a sub-sample of parents from our larger sample of parents, and 10 clinicians. The findings will inform the final protocol for a larger, efficacy trial.

ELIGIBILITY:
Inclusion Criteria Parents:

* Reside in the United States or one of its recognized territories
* Conceived 1 or more children via gamete (egg/sperm) or embryo donation who are currently between the ages of 1 - 16 years of age
* Have not informed their child(ren) about their donor conception origins
* Are 21 years-of-age or older
* English speaking

Inclusion Criteria Clinicians:

* Active practice as a healthcare professional (e.g., nurse, physician, psychologist, social worker)
* Provide education and/or counseling to gamete (eggs, sperm) and/or embryo donation recipient parents about disclosure to their children in the United States or one of its recognized territories
* Able to provide feedback and insight about new tools to assist gamete (eggs, sperm) and/or embryo donation recipient parents with disclosure to their donor-conceived children
* Are 21 years-of-age or older
* English speaking

Exclusion Criteria Parents:

* Have already disclosed the donor conception to their donor-conceived child or children
* Reside outside of the United States or one of its recognized territories

Exclusion Criteria Clinicians:

* Not directly involved in providing education and/or counseling to gamete (eggs, sperm) and/or embryo donation recipient parents about disclosure to their children
* Are a member of the research team

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Hershberger, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
When we publish our results, electronic copies of publications will be deposited in PubMed Central within four weeks of acceptance by a journal. We will also submit our results to ClinicalTrials.gov Protocol Registration and Results System as required.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TELL Tool Group | eBook Attention-Control
Started | 41 | 34
Recruitment Goal Achieved | 41 | 34
Completed | 30 | 30
Not Completed | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TELL Tool Group | eBook Attention-Control | Total
Number analyzed (Participants) | 41 | 34 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 34 | 75
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 31 | 70
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 36 | 30 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 35 | 30 | 65
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 34 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Disclosed the Donor Conception to Their Children
Description: Participant's report of current state of disclosure to their child or children. Total score range = 1 (disclosed) 2 (not-disclosed)
Time Frame: Disclosure assessed at 4-week time point. Data for the 12-week time point was missing due to a technology issue.
Measure: Count of Participants; unit: Participants
Arm/Group | TELL Tool Group | eBook Attention-Control
Number analyzed (Participants) | 30 | 30
Participants | 23 | 16

2. Secondary Outcome: Change in Disclosure Intention
Description: Parent's report on the Survey about Parents' Disclosure Intention. No score range (13 items)
Time Frame: Baseline-Change in Disclosure Intention at Immediate posttest-Month 1-Month 3
Reporting Status: Not Posted

3. Secondary Outcome: Change in Disclosure Competence
Description: Parent's report on the Perceived Competence Scale. Total score range = 4 (worse) to 28 (better)
Time Frame: Baseline-Change in Disclosure Competence at Immediate posttest-Month 1-Month 3
Reporting Status: Not Posted

4. Secondary Outcome: Change in Disclosure Anxiety
Description: Parent's report on the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety - Computer Adapted Test (CAT). Total scores for CAT will be comparable across participants.
Time Frame: Baseline-Change in Disclosure Anxiety at Immediate posttest-Month 1-Month 3
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Acceptability of the TELL Tool and eBook
Description: Participant's reports to the Acceptability Survey. No score range (19 items)
Time Frame: Immediate posttest
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Acceptability of the TELL Tool, eBook and Study Protocol
Description: Participant's responses to the Cognitive Interviews. No score range (Cognitive Interview Guide for Acceptability)
Time Frame: Month 15
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pretesting of the Measures
Description: Participant's (8 to 12 participants who are not part of the pilot randomized controlled trial) responses to Cognitive Interviews. No score range. (Cognitive Interview Guide for Measures)
Time Frame: Before baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Parents who participated in the pilot, RCT were assessed about adverse events at the 4-week and 12-week post-test data collection time points. The overall implementation of the pilot, RCT was from recruitment of our first parent participant into the pilot, RCT on July 26, 2021 through the 12-week post-test time point, which was September 30, 2022 when data collection for the pilot, RCT was completed.
Description: At the conclusion of the 4-week and 12-week data collection time points, participants were asked via an open-ended survey question about their reaction to participating in the study to assess for adverse events. For parents that reported disclosure to their children at the 4-week or 12-week time points, parent participants were asked about their child(ren)'s reaction(s) to the disclosure.
Arm/Group | TELL Tool Group | eBook Attention-Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/34
Other Adverse Events (participants affected / at risk) | 0/41 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04841967/Prot_SAP_000.pdf